CLINICAL TRIAL: NCT04963764
Title: Procalcitonin to Reduce Antibiotic Use in Pediatric Pneumonia
Acronym: PRAPP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Children's Hospital of Philadelphia (Other); Children's Hospital Medical Center, Cincinnati (Other); University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 1R34HL153474-01 (NIH)
Record Dates: First submitted 2021-06-16; First posted 2021-07-15 (Actual); Results first posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2022-10

CONDITIONS: Pneumonia; Pediatric Respiratory Diseases; Antibiotic Use; Community-acquired Pneumonia
Keywords: Pediatrics; Pediatric CAP; Pediatric Pneumonia; Antibiotic Use
MeSH Terms: conditions — Pneumonia; Community-Acquired Pneumonia | interventions — Amoxicillin

STUDY DESIGN:
Intervention Model Description: Pilot Feasibility Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Randomization to receive either oral placebo or amoxicillin for a standard course (10 days)
  Interventions: Drug: Placebo
- Amoxicillin (Active Comparator): Randomization to receive either oral amoxicillin or placebo for a standard course (10 days)
  Interventions: Drug: Amoxicillin

INTERVENTIONS:
Drug: Amoxicillin — Participants will be randomized to receive oral amoxicillin for a standard course (10 days)
  Arms: Amoxicillin
Drug: Placebo — Participants will be randomized to receive oral placebo for a standard course (10 days)
  Arms: Placebo

SUMMARY:
This pilot study will evaluate study processes and feasibility of a future large-scale clinical trial that proposes to test whether low-risk children managed as outpatients with community-acquired pneumonia (CAP) and procalcitonin (PCT) levels <0.25 ng/mL treated with placebo have a similar clinical response to those treated with antibiotics and fewer adverse effects.

DETAILED DESCRIPTION:
This pilot clinical trial is a 3-site, randomized, placebo-controlled, double-blinded trial assessing the feasibility of comparing amoxicillin to placebo in children 12 months to <6 years of age who present to the ED with Community Acquired Pneumonia (CAP), a procalcitonin (PCT) concentration of <0.25 ng/mL, and who will be treated as outpatients.

Screening and Enrollment This pilot feasibility trial will enroll over a 6-month period and take place at three sites (Ann and Robert H. Lurie Children's Hospital of Chicago, Cincinnati Children's Hospital Medical Center and The Children's Hospital of Philadelphia) that are or were members of the Pediatric Emergency Care Applied Research Network (PECARN). This study aims to enroll 36 patients in total (2 patients per month, per site). Clinical research coordinators (CRCs) at participating EDs will screen potentially eligible patients with respiratory tract symptoms and discuss eligibility with the treating attending physician. If thought to be eligible and a diagnosis of CAP is presumed by the treating physician, the CRC will approach the patient to complete screening procedures. The study will proceed in 2 stages, each with its own informed consent process. During Stage 1, baseline characteristics and serum PCT levels will be ascertained. Stage 2 will consist of a randomized trial of amoxicillin vs. placebo in the subset of patients from Stage 1 that have PCT <0.25 ng/mL.

Randomization After enrollment and confirmation of a PCT <0.25 ng/mL, patients will be randomized to a 10-day course of either amoxicillin (80-100 mg/kg divided BID up to 4,000 mg/day) or placebo. Randomization to amoxicillin or placebo will be at a 1:1 ratio with block sizes of 2 and 4. Patients will be stratified by the clinical site and randomization will be performed through an online system. As a double-blind clinical trial, the study patients and their parents/guardians, investigators and study staff will be blinded to study treatment assignment for the duration of the study.

Study Drug Administration Local investigational drug pharmacies will be provided with active study medication (i.e., amoxicillin) and matching placebo. Site pharmacies at each institution will store study drug and dispense as needed. Study medications will both be liquid reconstituted from powder, and will resemble each other with regards to appearance, favor, consistency and packaging. Study products will be labeled with numerical codes that will maintain allocation concealment. Site investigational pharmacies will be provided with amoxicillin and placebo, in addition to the randomization scheme. The pharmacy will aliquot amoxicillin and placebo into blinded bottles based on randomization scheme.

Follow-up The guardians of participants will be asked to complete a daily symptom diary, using an online data collection form in REDCap, during the first 7 days after the initial Emergency Department study visit. The follow-up will assess patient condition, clinical response, signs or symptoms of clinical deterioration and other adverse effects. The primary outcome will be assessed at day 7 (+/- 2 days), using video chat technology that is standard on most smart phones, tablets, and computers. Video follow-up will be performed by site clinician investigators. In the rare case that a mobile device or computer with video chat technology is not available to the family, the day 7 follow-up will occur by telephone or text through an online system. A final follow-up, performed by site research staff, by telephone call, will occur at Day 21 (+/- 2 days) to assess overall disease course and secondary outcomes.

Data Collection At baseline, demographics, medical history, and history of current illness will be obtained from all participants during stage 1 (pre-randomization). Vital signs will be obtained and a brief physical examination will be performed. After the initial ED visit, patients will record symptoms on daily basis for 6 days via an online data collection form. Follow-up assessments will be completed via telehealth visit or telephone for days 7 and 21. Follow-up visits will collect data regarding symptoms, adverse events and return to medical care, in addition to assessing adherence to study procedures (i.e., medication adherence and daily symptom diary completion). If there is concern for adverse events or deterioration that may warrant medical care, the participant's caregiver will be instructed to contact their primary care physician, emergency department, or call 911, as indicated.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12-71 months; and
2. Diagnosis of CAP, defined using established criteria:

   1. Signs and symptoms of lower respiratory tract infection (LRTI), defined as one or more of the following:

      * new or different cough; or
      * new or different sputum production; or
      * chest pain; or
      * dyspnea/shortness of breath; or
      * documented tachypnea; or
      * abnormal findings consistent with LRTI on physical examination (e.g., crackles/rales, rhonchi, wheezing) and
   2. Fever, defined as temperature greater than or equal to 38 degrees C, and
   3. ED clinician diagnosis of CAP, including intention to treat with antibiotics, and
   4. Chest radiography suspicious for CAP
3. Treatment as an outpatient after ED visit.
4. Procalcitonin < 0.25 ng/mL

Exclusion Criteria:

1. Hospitalization within 7 days preceding study visit; or
2. Sustained oxygen saturations <90% with appropriate waveform on oximeter; or
3. Incomplete immunization status (<3 doses of Hib and pneumococcal vaccines; or
4. Chronic complex medical conditions (chronic heart disease, chronic lung disease (not including asthma), congenital airway or lung malformations, cystic fibrosis, chronic renal disease, protein-losing enteropathy, genetic syndromes, neurocognitive deficits, or metabolic disorders); or
5. Conditions that compromise the immune system (HIV, primary immunodeciency, asplenia, sickle cell disease, receipt of hematopoietic stem cell or solid organ trans- plant, immunosuppressive agents, daily corticosteroids for more than 7 consecutive days in past 14 days) ; or
6. Systemic antibiotic receipt within the previous 7 days of CAP diagnosis; or
7. Radiographic findings of complicated pneumonia (moderate-to-large pleural effusion, empyema, abscess, necrotic lung disease) ; or
8. Pneumonia known to be due to bacterial source at the time of enrollment, as documented by blood culture or PCR if available, or another clear source of bacterial infection requiring immediate antibiotics; or
9. Toxic clinical appearance, sepsis, or critical illness as determined by clinical team at ED presentation; or
10. Diagnosed with pneumonia in previous 6 months; or
11. Provider diagnosis of bronchiolitis, bronchitis, or aspiration pneumonia; or
12. Concomitant asthma exacerbation requiring systemic corticosteroids; or
13. Severe drug allergy to amoxicillin; or
14. Any other condition that in the judgement of investigators or the clinical team could affect safety of the subject; or
15. No access to a telephone or video technology for follow-up; or
16. Current enrollment in another clinical trial of an investigational agent; or
17. Previous enrollment in this trial.

Ages: 12 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-05-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
The P-RAPP research team and the PECARN Data Coordinating Center (DCC) at the University of Utah is committed to publicly sharing data for each trial in which we participate in compliance with the NIH's data-sharing policy. As this is a pilot study, a public use dataset will not be developed.

RESULTS

PARTICIPANT FLOW:
Groups:
- Stage 1 - Consented to Have Procalcitonin Testing Performed: Enrolled participants with procalcitonin testing performed
- Stage 2 - Placebo: Randomization to receive either oral placebo or amoxicillin for a standard course (10 days)
  Placebo: Participants will be randomized to receive oral placebo for a standard course (10 days)
- Stage 2 - Amoxicillin: Randomization to receive either oral amoxicillin or placebo for a standard course (10 days)
  Amoxicillin: Participants will be randomized to receive oral amoxicillin for a standard course (10 days)
Period: Stage 1
Arm/Group | Stage 1 - Consented to Have Procalcitonin Testing Performed | Stage 2 - Placebo | Stage 2 - Amoxicillin
Started | 5 | 0 (Enrollment in the Stage 2 - Placebo Arm did not apply to Stage 1 of the study.) | 0 (Enrollment in the Stage 2 - Amoxicillin Arm did not apply to Stage 1 of the study.)
Completed | 5 | 0 (Enrollment in the Stage 2 - Placebo Arm did not apply to Stage 1 of the study.) | 0 (Enrollment in the Stage 2 - Amoxicillin Arm did not apply to Stage 1 of the study.)
Not Completed | 0 | 0 | 0
Period: Stage 2
Arm/Group | Stage 1 - Consented to Have Procalcitonin Testing Performed | Stage 2 - Placebo | Stage 2 - Amoxicillin
Started | 0 (Enrollment in the Stage 1 - Consented to have Procalcitonin Testing Performed Arm did not apply to Stage 2 of the study.) | 0 (No participants were enrolled in the Stage 2 - Placebo Arm.) | 1
Completed | 0 (Enrollment in the Placebo Arm did not apply to Stage 1 of the study.) | 0 (No participants were enrolled in the Stage 2 - Placebo Arm.) | 0
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline data only collected for Stage 2.
  No participants were enrolled in the Stage 2 - Placebo Arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage 2 - Placebo | Stage 2 - Amoxicillin | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Customized [Count of Participants; unit: Participants]
  Age 12-71 Months | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Total Pilot Trial Enrollment
Description: Number of patients enrolled in Stage 2 (Randomized Pilot Trial) per site
Time Frame: Day 7
Population: The one participant in the Amoxicillin arm withdrew from the study on Day 7. There were no participants enrolled in the Placebo arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Amoxicillin
Number analyzed (Participants) | 0 | 1
Participants | 0 | 1

2. Secondary Outcome: Consent Rate for Stage 1 (Procalcitonin Ascertainment)
Description: Number of eligible participants approached regarding trial participation who provided informed consent to participate in Stage 1 of the trial compared with number of participants approached for participation
Time Frame: Measured at completion of pilot trial (6 months)
Population: Of 36 eligible participants approached, five (13.9%) provided informed consent to be included in Stage 1
Measure: Count of Participants; unit: Participants
Groups:
- Percentage of Eligible Participants Approached Who Consented for Inclusion in Stage 1: Number of Eligible Participants Approached Who Provided Informed Consent in Stage 1/Number of participants approached for participation
Arm/Group | Percentage of Eligible Participants Approached Who Consented for Inclusion in Stage 1
Number analyzed (Participants) | 36
Participants | 5

3. Secondary Outcome: Rate of Eligible Participants for Stage 2 (Randomized Pilot Trial)
Description: Proportion of participants who received procalcitonin in Stage 1 who had an eligible procalcitonin for Stage 2 (PCT <0.25)
Time Frame: Measured at completion of pilot trial (6 months)
Population: Of 5 eligible participants who received procalcitonin in Stage 1, 3 (60%) had PCT <0.25.
Measure: Count of Participants; unit: Participants
Groups:
- Rate of Eligible Participants for Stage 2: Proportion of participants who received procalcitonin in Stage 1 who had an eligible procalcitonin for Stage 2 (PCT <0.25)
Arm/Group | Rate of Eligible Participants for Stage 2
Number analyzed (Participants) | 5
Participants | 3

4. Secondary Outcome: Consent Rate for Stage 2 (Randomized Pilot Trial)
Description: Number of eligible participants for Stage 2 (PCT <0.25) who provided informed consent to participate in Stage 2 of the trial compared with number of eligible participants approached for participation
Time Frame: Measured at completion of pilot trial (6 months)
Population: Of the 2 eligible participants for Stage 2 who were approached, one provided informed consent for Stage 2.
Measure: Count of Participants; unit: Participants
Groups:
- Consent Rate for Stage 2 (Randomized Pilot Trial): Number of eligible participants for Stage 2 (PCT <0.25) who provided informed consent to participate in Stage 2 of the trial compared with number of eligible participants approached for participation
Arm/Group | Consent Rate for Stage 2 (Randomized Pilot Trial)
Number analyzed (Participants) | 2
Participants | 1

5. Secondary Outcome: Lost to Follow-Up at Day 7
Description: Number of enrolled participants who did not complete the Day 7 follow-up visit
Time Frame: Day 7
Population: No patients were randomized to the Placebo group. One patient withdrew from the Amoxicillin group on Day 7. Therefore, this patient was lost to follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Amoxicillin
Number analyzed (Participants) | 0 | 1
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data was tracked through Day 7.
Description: Adverse events were only monitored during Stage 2.
  The one enrolled patient withdrew at Day 7 and did not report any adverse events up until that time point.
Arm/Group | Stage 2 - Placebo | Stage 2 - Amoxicillin
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

LIMITATIONS AND CAVEATS:
Enrollment occurred during the COVID-19 pandemic when pediatric pneumonia numbers were lower than current (and pre-pandemic) numbers, which significantly affected enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/64/NCT04963764/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-05): https://cdn.clinicaltrials.gov/large-docs/64/NCT04963764/SAP_001.pdf